CLINICAL TRIAL: NCT01656850
Title: The Effect of Whole Almonds on Glucoregulation, Endothelial Function, Inflammation, Lipid Profile, and Oxidative Stress in Chinese Patients With Type 2 Diabetes
Brief Title: The Effect of Whole Almonds on Biomarkers of Cardiovascular Disease in Chinese Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Jen-Fang Liu, Professor, Taipei Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PV0805
Record Dates: First submitted 2012-01-13; First posted 2012-08-03 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
Keywords: hyperglycemia; hyperinsulinemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Almond diet first, then NCEP Diet (Experimental): In a 28-wk randomized, cross-over, controlled feeding trial with a 2 week washout between alternative diets, subjects were assigned to receive NCEP or almond diet for 12 weeks after a 2-weeks run-in period
  Interventions: Other: Almond diet first, then NCEP Diet
- NCEP diet first, then Almond diet (Experimental): In a 28-wk randomized, cross-over, controlled feeding trial with a 2 week washout between alternative diets, subjects were assigned to receive NCEP or almond diet for 12 weeks after a 2-weeks run-in period
  Interventions: Other: NCEP diet first, then Almond diet

INTERVENTIONS:
Other: Almond diet first, then NCEP Diet — whole almonds will be incorporated into a control diet which is a NCEP step 2 diet. Whole almonds will replace 20% daily calorie intake. Subjects were assigned to receive almond diet for 12 weeks after a 2-weeks run-in period. After washout 2 weeks, change diet to NCEP Diet for 12 weeks
  Arms: Almond diet first, then NCEP Diet
Other: NCEP diet first, then Almond diet — NCEP diet first, then Almond diet. Subjects were assigned to receive NCEP diet for 12 weeks after a 2-weeks run-in period. After washout 2 weeks, change diet to almond diet for 12 weeks
  Arms: NCEP diet first, then Almond diet

SUMMARY:
The purpose of the study is to examine whether almond consumption for 3 month will help Chinese patients with type 2 diabetes control blood glucose and decrease risk factors of cardiovascular disease.

DETAILED DESCRIPTION:
Our previous study demonstrated almonds (~60 g/d) improved lipid profile, glucoregulation, inflammation, and oxidative stress in 20 Chinese patients with type 2 diabetes mellitus (T2DM). To follow-up and expand this work with a more robust trial, the investigators propose a larger (n = 40), longer-term (90-d) investigation of the effect of almonds (~60 g/d) on adipokine regulation, endothelial function, glucoregulation, inflammation, lipid profile, and oxidative stress in Chinese patients with T2DM as compared to a placebo control. The investigators will conduct a 7-mo randomized, cross-over, placebo controlled clinical trial in which all meals will be provided to all subjects (n = 40). During the first 2 weeks (run-in period), all subjects will receive a control diet resembling a typical Taiwan diet, prepared based on the NCEP Step 2 guidelines. During the following 3 mo (Phase I), subjects will be randomized to receive either the control diet or the control diet with whole almonds (~60g/d) incorporated to replace 20% calories. After a 2-wk washout period during which all subjects will once again receive the control diet, subjects will receive the opposite diet to the one assigned during the Phase I for the other 3 months (Phase II). The caloric content of each diet will be adjusted to each subjects' energy needs to prevent any change in body weight. The following biomarkers will be determined at the baseline and end of each dietary intervention: Glucoregulation: fasted serum HbA1c, glucose and insulin, postprandial serum glucose and insulin, and urinary C-peptide; Endothelial Function: brachial artery FMD and serum nitric oxide, e-selectin, endothelial-1 (ET-1), and intracellular adhesion molecule-1 (ICAM-1); Adipokine Regulation: serum adiponectin, leptin, and resistin; Inflammation: serum high-sensitivity C-reactive protein (CRP), interleukin (IL)-6, IL-10, retinol binding protein-4 (RBP-4), and tumor necrosis factor (TNF)-α; Oxidative Stress: urinary isoprostanes (adjusted for creatinine) and serum protein carbonyls and oxidized LDL; and Lipid Profile: serum cholesterol, triglycerides, and apolipoproteins A1 and B.

ELIGIBILITY:
Inclusion Criteria:

* aged between 40-70 years,
* with BMI = 24-35 kg/m2,
* HbA1c 6.5-9 %, and
* regular use of oral hypoglycemic agents.

Exclusion Criteria:

* Use of insulin to control blood glucose
* Regular use of oral steroids
* Regular use of anti-inflammatory agents (prescribed [Rx] or over-the-counter [OTC])
* Gain or loss of larger than 5% of body weight in the last 6 months
* CVD: coronary artery disease, left ventricular hypertrophy evidenced by echocardiogram, congestive heart failure, cerebrovascular disease, stroke, peripheral vascular disease, dysautonomia
* Gastrointestinal: diseases, conditions, or medications influencing gastrointestinal absorption including active peptic ulcer disease, inflammatory bowel disease, treatment with acid-lowering drugs
* Renal: chronic kidney disease due to any condition, renovascular disease, history of nephrolithiasis, diabetic nephropathy, serum creatinine > 1.5 mg/dL
* Endocrine: disease, untreated thyroid disease, adrenal disease, pheochromocytoma, parathyroid disease, hyperuricemia
* Rheumatologic: gout, inflammatory arthritis
* Active treatment for cancer of any type (except basal cell carcinoma) 1 year
* Systolic blood pressure larger than 150 mmHg, and diastolic blood pressure larger than 95 mmHg.
* Any history of or known allergies to nuts of any kind
* Frequent nut consumption, defined as ≥ 3 oz/wk; however, subjects who are willing to refrain from eating all nuts and nut products for 6 wk prior to their initial visit (Visit 1) may be considered eligible
* Regular use of any dietary supplements containing vitamins, minerals, herbal or other plant-based preparations, fish oil supplements (including cod liver oil) or homeopathic remedies; however, subjects who are willing to refrain from the use of these supplements for 1 mo prior to their initial visit (Visit 1) and throughout the entire study may be considered eligible
* Usual daily ethanol intake of larger or equal to 2 drinks (24 oz beer, 8 oz wine, 2 oz hard liquor)
* Illicit drug use
* Specific laboratory blood or urine analysis parameters of: creatinine larger than 1.5 mg/dL, ALT and AST larger than 1.5 nmol/L, and urinalysis - hematuria and proteinuria

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Fang Liu, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen CM, Liu JF, Li SC, Huang CL, Hsirh AT, Weng SF, Chang ML, Li HT, Mohn E, Chen CO. Almonds ameliorate glycemic control in Chinese patients with better controlled type 2 diabetes: a randomized, crossover, controlled feeding trial. Nutr Metab (Lond). 2017 Aug 2;14:51. doi: 10.1186/s12986-017-0205-3. eCollection 2017. PMID 28785295

RESULTS

PARTICIPANT FLOW:
Groups:
- Whole Almonds First, Then NCEP Diet: run in 2 weeks, whole almonds diet Intervention (3 months), Washout (2 weeks), and then NCEP diet Intervention (3 months)
- NCEP Diet First, Then Whole Almonds Diet: run in 2 weeks, NCEP diet Intervention (3 months), Washout (2 weeks), whole almonds Intervention (3 months)
Period: First Intervention (3 Months)
Arm/Group | Whole Almonds First, Then NCEP Diet | NCEP Diet First, Then Whole Almonds Diet
Started | 20 | 20
Completed | 17 | 16
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4
Period: Washout (2 Weeks)
Arm/Group | Whole Almonds First, Then NCEP Diet | NCEP Diet First, Then Whole Almonds Diet
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Second Intervention (3 Months)
Arm/Group | Whole Almonds First, Then NCEP Diet | NCEP Diet First, Then Whole Almonds Diet
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Almond Diet First, Then NCEP Diet: whole almonds to replace 20% daily calorie intake
  whole almonds: Whole almonds will be incorporated into a control diet which is a NCEP step 2 diet. Whole almonds will replace 20% daily calorie intake.
- NCEP Diet First, Then Almond Diet: follow NCEP step 2 diet
  NCEP Step 2 diet: follow NCEP step 2 diet
- Total: Total of all reporting groups
Arm/Group | Almond Diet First, Then NCEP Diet | NCEP Diet First, Then Almond Diet | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 4 | 2 | 6
Gender [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  Taiwan | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Major Nutrients of NCEP Step 2 Diet and Almond Diets
Time Frame: the entire study, up to 3 months
Measure: Mean (Standard Deviation); unit: % of energy
Groups:
- Whole Almonds: whole almonds to replace 20% daily calorie intake
  whole almonds: Whole almonds will be incorporated into a control diet which is a NCEP step 2 diet. Whole almonds will replace 20% daily calorie intake.
- NCEP Step 2 Diet: follow NCEP step 2 diet
  NCEP Step 2 diet: follow NCEP step 2 diet
Arm/Group | Whole Almonds | NCEP Step 2 Diet
Number analyzed (Participants) | 33 | 33
% of energy
  Crude protein | 17.5 (1.3) | 17.2 (1.6)
  Fat | 38.4 (3.5) | 29.2 (3.1)
  Carbohydrate | 47.0 (3.4) | 55.7 (4.3)
Statistical Analysis 1: Comparison: Whole Almonds vs NCEP Step 2 Diet; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

2. Primary Outcome: Plasma Lipid Profiles at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Con Before: before consuming NCEP step II diet
- Con After: after consuming NCEP step II diet for 3 months
- Alm Before: before consuming almond diet
- Alm After: after consuming almond diet for 3 months
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
mg/dL
  HDL | 44.8 (12.9) | 49.7 (13.4) | 45.2 (11.9) | 48.5 (12.4)
  LDL | 97.5 (29.3) | 102.9 (29.2) | 100.2 (29.5) | 98.0 (24.5)
  Total cholesterol | 170.7 (31.9) | 180.6 (36.0) | 175.1 (36.0) | 178.9 (28.4)
  Triglyceride | 161.1 (83.7) | 141.2 (68.3) | 175.1 (36.0) | 178.9 (28.4)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.2786, Mixed Models Analysis

3. Primary Outcome: The Calories of NCEP Step 2 Diet and Almond Diets
Time Frame: the entire study, up to 3 months
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Whole Almonds | NCEP Step 2 Diet
Number analyzed (Participants) | 33 | 33
kcal | 1,665.9 (153.8) | 1,643.4 (133.6)
Statistical Analysis 1: Comparison: Whole Almonds vs NCEP Step 2 Diet; Test type: Superiority or Other; p = 0.420, Mixed Models Analysis

4. Primary Outcome: Lipid Composition of NCEP Step 2 Diet and Almond Diets
Time Frame: the entire study, up to 3 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Whole Almonds | NCEP Step 2 Diet
Number analyzed (Participants) | 33 | 33
g
  PUFA | 22.0 (4.1) | 22.3 (4.5)
  MUFA | 30.7 (4.0) | 12.7 (3.3)
  SFA | 11.1 (3.3) | 9.5 (2.6)
Statistical Analysis 1: Comparison: Whole Almonds vs NCEP Step 2 Diet; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

5. Primary Outcome: Body Weight at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
kg | 64.7 (10.8) | 64.8 (11.0) | 65.3 (11.0) | 64.7 (10.7)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.2412, Mixed Models Analysis

6. Primary Outcome: Body Fat Percentage at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
percentage of body weight | 31.6 (8.73) | 31.4 (9.40) | 31.0 (8.95) | 31.7 (8.63)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.3837, Mixed Models Analysis

7. Primary Outcome: Blood Pressure at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
mmHg
  SBP | 124.2 (15.2) | 123.6 (18.2) | 124.5 (14.0) | 122.1 (13.4)
  DBP | 74.9 (10.3) | 77.3 (9.84) | 74.9 (10.6) | 76.5 (10.2)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.9784, Mixed Models Analysis

8. Primary Outcome: Plasma Fasting Glucose at the Baseline and the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
mg/dL | 146.5 (37.9) | 139.6 (33.1) | 140.7 (30.9) | 140.3 (36.8)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.5868, Mixed Models Analysis

9. Primary Outcome: Area Under Curve of Plasma Glucose After Eating Standard Breakfast at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: mg.min/dL
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
mg.min/dL | 37424 (7681) | 36415 (7250) | 35768 (7379) | 37706 (8490)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.1101, Mixed Models Analysis

10. Primary Outcome: Plasma Fasting Insulin at the Baseline and the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
mU/L | 11.2 (4.9) | 12.3 (6.0) | 10.4 (4.6) | 11.8 (5.7)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.7823, Mixed Models Analysis

11. Primary Outcome: Area Under Curve of Plasma Insulin After Eating Standard Breakfast at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: mU.min/L
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
mU.min/L | 3975 (2353) | 4690 (3327) | 4055 (2964) | 4345 (2791)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.5570, Mixed Models Analysis

12. Primary Outcome: Plasma HbA1c Level at the Baseline and the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: percentage of hemoglubin
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
percentage of hemoglubin | 7.47 (1.12) | 7.45 (0.80) | 7.51 (0.97) | 7.39 (1.05)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.6263, Mixed Models Analysis

13. Primary Outcome: HOMA at the Baseline and the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
pg/mL | 4.00 (2.08) | 4.24 (2.70) | 3.58 (1.75) | 3.98 (1.98)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.8328, Mixed Models Analysis

14. Primary Outcome: Plasma Apolipoprotein Level at the Baseline and the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
g/L
  Apo A1 | 128.9 (23.9) | 135.1 (23.4) | 128.3 (22.8) | 135.3 (24.3)
  Apo B | 82.9 (22.2) | 85.8 (24.2) | 84.3 (23.3) | 86.7 (22.6)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.7758, Mixed Models Analysis

15. Primary Outcome: Plasma Nitric Oxide Level at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
μmol/L | 59.6 (35.8) | 72.1 (55.3) | 62.5 (40.9) | 50.6 (26.7)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.0476, Mixed Models Analysis

16. Primary Outcome: Endothelial Function at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
ng/mL
  sE-Selectin | 43.4 (20.7) | 44.0 (20.2) | 46.1 (18.0) | 42.3 (15.5)
  ICAM-1 | 22.3 (7.74) | 22.9 (7.22) | 24.0 (8.91) | 23.1 (8.09)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.1205, Mixed Models Analysis

17. Primary Outcome: Plasma Protein Carbonyl Level at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: nmol/mg
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
nmol/mg | 1.00 (0.54) | 1.06 (0.68) | 1.00 (0.65) | 0.72 (0.56)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.1512, Mixed Models Analysis

18. Primary Outcome: Plasma Oxide LDL Level at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
U/L | 32.8 (9.9) | 34.8 (10.9) | 33.9 (10.9) | 35.1 (9.9)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.7364, Mixed Models Analysis

19. Primary Outcome: Urine Isoproterenol Level at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
ng/mg creatinine | 12.2 (6.19) | 14.2 (9.22) | 11.9 (4.24) | 12.2 (4.68)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.1995, Mixed Models Analysis

20. Primary Outcome: Plasma Vitamin E Level at the Baseline and at the End of 3-month Dietary Intervention
Time Frame: at the baseline and at the end of 3-month dietary intervention
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Con Before | Con After | Alm Before | Alm After
Number analyzed (Participants) | 33 | 33 | 33 | 33
μmol/L | 8.51 (3.37) | 9.24 (5.45) | 8.86 (4.43) | 9.57 (5.11)
Statistical Analysis 1: Comparison: Con Before vs Con After vs Alm Before vs Alm After; Test type: Superiority or Other; p = 0.8528, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: one week for each intervention
Groups:
- Whole Almond Diet: participants received experiment diet containing 20% calorie from whole almond
- NCEP Diet: participants received NCEP diet for 3 months
Arm/Group | Whole Almond Diet | NCEP Diet
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No